CLINICAL TRIAL: NCT02215603
Title: Effects of Disrupting Prolonged Sitting With Different Physical Activity Protocols on Metabolic Risk Factors in Sedentary Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ProlongedSitting
Record Dates: First submitted 2014-08-07; First posted 2014-08-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Prolonged Sitting; Breaking Prolonged Sitting With Physical Activity
MeSH Terms: interventions — Exercise

ARMS (4):
- Prolonged sitting (No Intervention): 9 h of prolonged sitting
- Prolonged sitting + interval standing bouts (Experimental): Stand bout for 15-min every 30 minutes during the 9 hours of sitting
  Interventions: Behavioral: Breaking prolonged sitting with physical activity
- Moderate exercise bout + Prolonged sitting (Experimental): 30-min moderate-intensity exercise bout followed by 8 h of sitting
  Interventions: Behavioral: Breaking prolonged sitting with physical activity
- Moderate exercise bout + Prolonged sitting +Standing bouts (Experimental): 30-min moderate-intensity exercise bout and stand bout for 15-min every 30 minutes during the remaining 8 hours of sitting
  Interventions: Behavioral: Breaking prolonged sitting with physical activity

INTERVENTIONS:
Behavioral: Breaking prolonged sitting with physical activity
  Arms: Moderate exercise bout + Prolonged sitting; Moderate exercise bout + Prolonged sitting +Standing bouts; Prolonged sitting + interval standing bouts

SUMMARY:
Great controversy exists with respect to the optimal or the minimum volume, intensity, and frequency of physical activity capable of attenuating the hazards of prolonged sitting on the metabolic profile. Thus, our study aims to comprehensively investigate the effects of disrupting prolonged sitting with different physical activity protocols on metabolic risk factors in sedentary males.

Ten sedentary males will take part in this randomized cross-over trial consisting of four 27-h conditions. All conditions will be identical except for the physical activity: prolonged sitting intervention (SIT) participants will sit continuously for 9 hours; prolonged sitting+interval standing intervention (STAND), participants will stand for 15 min every 30 minutes (total 270 min) during the 9 hours of sitting; prolonged sitting+moderate-intensity exercise bout (MVPA) participants will perform a 30-min moderate-intensity exercise bout on a treadmill (energy-matched to STAND), after which they will sit for the remaining time; and prolonged sitting+moderate-intensity exercise bout +interval standing intervention (MVPA-STAND), participants will perform a 30-min moderate-intensity exercise bout on a treadmill (energy-matched to STAND), after which they will stand for 15 min every 30 minutes (total 240 min) during the remaining 8 hours of sitting. Blood glucose, insulin, lipids and cytokines will be determined.

The investigators expect that disrupting prolonged sitting with intermittent standing and a moderate-exercise bout will positively affect the metabolic profile of the participants. Furthermore, we will investigate if combined, these strategies will have an additive effect.

ELIGIBILITY:
Inclusion Criteria:

* Males,
* age 25-55 y,
* BMI >18 and <35 kg/m2

Exclusion Criteria:

* Clinically diagnosed diabetes,
* dyslipidaemia,
* hypertension,
* use of glucose- and/or lipid-lowering medication,
* smoking,
* evidence of thyroid, liver, lung, heart or kidney disease,
* non-sedentary occupation and primary means of commuting to work (i.e., cycling) in the last 4 months,
* VO2max levels above the considered average fitness according to age,
* contraindication to increased levels of physical activity.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of glucose and insulin postprandial responses | 27 h
  Glucose and insulin levels will be assessed 10 min before, and 30, 60, 120 and 180 min after each main meal. These postprandial responses will be defined as the area under the curve (AUC) assessed over the 3-h period after each main meal (3-h AUC) and the cumulative AUC after all main meals (12-h AUC).

SECONDARY OUTCOMES:
Glucose levels | 27 hours
  Glucose incursions will measured using the glucose monitoring (CGM) system throughout the 27 hours. Mean, maximum and minimum glucose values during the 27h will be the outcome measures (mmol/l).
Area under the curve of lipid postprandial responses | 27 h
  Lipid levels will be assessed 10 min before, and 30, 60, 120 and 180 min after each main meal. These postprandial responses will be defined as the area under the curve (AUC) assessed over the 3-h period after each main meal (3-h AUC) and the cumulative AUC after all main meals (12-h AUC).

OTHER OUTCOMES:
Area under the curve of cytokine postprandial responses | 27 h
  Cytokine levels (TNF-alpha, IL-6, IL-10, and IL1-ra) will be assessed 10 min before, and 30, 60, 120 and 180 min after each main meal. These postprandial responses will be defined as the area under the curve (AUC) assessed over the 3-h period after each main meal (3-h AUC) and the cumulative AUC after all main meals (12-h AUC).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Inflammation and Metabolism, Copenhagen, Denmark